CLINICAL TRIAL: NCT06356545
Title: A Case-control Study of Phenotype and Multi-omics Analysis of Children With Congenital Diarrhea and Enteropathy in China
Brief Title: Phenotype and Multi-omics Analysis of Children With Congenital Diarrhea and Enteropathy in China
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: OMICS_CODE_01
Record Dates: First submitted 2024-03-21; First posted 2024-04-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diarrhea Infantile
MeSH Terms: conditions — Diarrhea, Infantile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Congenital diarrhea and enteropathy (CODE) patients
- Control: Healthy children

SUMMARY:
This study will establish a clinical cohort of children with congenital diarrhea and enteropathy (CODE), mine biomarkers of CODE through multi-omics technology and construct a clinical risk prediction model.

DETAILED DESCRIPTION:
This study will establish a clinical cohort and a clinical phenotype database of children with congenital diarrhea and enteropathy (CODE), The investigator will mine biomarkers of CODE through multi-omics technology. This study is designed to construct a clinical risk prediction model by combining artificial intelligence technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic diarrhea lasting greater than 2 months or greater than 1 month in patients younger than 2 months of age
* Patients with consent from parents or legal guardians

Exclusion Criteria:

* Chronic diarrhea caused by specific infections, i.e. CMV, Clostridioides difficile
* Chronic diarrhea with necrotizing enterocolitis, short bowel syndrome
* Functional diarrhea
* Patients with poor compliance

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with chronic diarrhea lasting greater than 2 months or greater than 1 month in patients younger than 2 months of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype of congenital diarrhea and enteropathy in China | Within approximately 2 years of enrollment
  Describe the clinical phenotype(Birth status, family history, clinical features of diarrhea, laboratory examination, endoscopic and histological evaluation results, growth and development indicators, previous treatment and effect were collected) of congenital diarrhea and enteropathy in China,We will use our own mobile application or to collect the relevant data, which will be filled in by the parents of the child.

SECONDARY OUTCOMES:
Biomarkers of congenital diarrhea and enteropathy with diagnostic value through microbiome, metabolome and proteome features | Within approximately 2 years of enrollment
  Plasma and stool were collected from patients and healthy control children for multi-omics screening to identify biomarkers, of which differential expression were mined through proteome(olink), microbiome(metagenomic sequencing) and metabolome( untargeted metabolomics)，relevant statistical analyses were performed using non-parametric tests, such as the Wilcoxon signed-rank test.
Cinical risk prediction model for congenital diarrhea and enteropathy built by artificial intelligence and machine learning | Within approximately 30 months of enrollment
  Using artificial intelligence and machine learning to construct predictive models for congenital diarrhea and enteropathy by combining children's clinical phenotypes and multi-omics results，such as the random forest model

CONTACTS AND LOCATIONS:
Locations (1):
- Yanqiu Wang, Shanghai, Shanghai Municipality, China